CLINICAL TRIAL: NCT07025317
Title: Developing an Evidence-based Approach to Diagnose and Treat Adults With a History of Concussion
Brief Title: Spotting and Managing Adult Repeated Traumas in the Brain
Acronym: SMARTBRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: University of Victoria (Other); NeuroTracker Athletics Inc. (Unknown); Brain Canada (Other); Consortium québécois sur la découverte du médicament (Unknown)
Responsible Party: Principal Investigator, Eduardo Lugo Arce, Coordinator, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Projet # 2024-5858; Faubert-SYN-347_NRFA (Other Grant/Funding Number: CQDM-BrainCanada-NeuroTracker)
Record Dates: First submitted 2025-05-05; First posted 2025-06-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Brain Injury Traumatic Mild
Keywords: Concussions; mild traumatic brain injury; mild brain traumas; NeuroTracker
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control lacks of perceptual-cognitive training (NeuroTracker) in individuals with and without prior mTBI.
- NeuroTracker (Experimental): NeuroTracker consists of perceptual-cognitive training in individuals with and without prior mTBI.
  Interventions: Other: Perceptual-cognitive

INTERVENTIONS:
Other: Perceptual-cognitive — The intervention is to determine the effectiveness of NeuroTracker for treating cognitive deficits associated with a prior history of concussion. NeuroTracker has a virtual cloud-based platform (NeuroTrackerX), which has been validated for use in research. This online platform allows participants to complete the interventions from home and greatly increases the accessibility of the program. Participants will have two 30-minute training sessions per week over the course of the 6-month intervention. Each session will consist of 3 blocks of 20 trials. For each trial in a block, participants sit upright, approximately 20" away from a standard computer or laptop screen, and wear anaglyph 3D glasses while focusing on the center of a standard 20" computer screen.
  Arms: NeuroTracker

SUMMARY:
Emerging evidence suggests that concussions (a type of mild traumatic brain injury; mTBIs) may cause chronic neurological disturbances with effects lasting beyond 20 years, changing brain structure and nearly doubling the risks of developing dementia into old age. Yet diagnoses remain notoriously difficult, gender differences are poorly understood, and negligible therapies exist to manage and treat these long-term effects.

This project proposes using a combination of NeuroTracker (a promising software-based cognitive assessment and intervention for mild TBIs), with the latest MRI techniques and blood-based biomarkers of brain function, to provide unprecedented assessment sensitivity of long-term concussion effects, comparing older male and female adults, with and without a history of concussion. Additionally, NeuroTracker will be used as a therapeutic intervention to improve outcomes in adults with histories of concussion, with the combined assessments measuring efficacy pre-post training.

This project aims to comprehensively understand the impacts of mild brain traumas into later life, via both physical and functional biomarkers of brain health. It will also validate the value of NeuroTracker as an accessible training intervention for recovering cognitive functions impacted by earlier-life concussions.

DETAILED DESCRIPTION:
Older adults with a history of concussions have a 2x greater risk of developing dementia, however it is not clear why some individuals show resilience and are cognitively healthy, while others struggle and show more pronounced cognitive deficits. Concussions are a form of mild traumatic brain injury (mTBI) that are induced by the impact of biomechanical forces on the brain. In Canada, there are approximately 94,000 activity-limiting concussions per year in individuals aged 12 and over (Statistics Canada). Despite increasing awareness of concussion risks, the objective assessment of long-term consequences of concussion remains a notoriously difficult clinical problem; a multimodal approach is required to improve the understanding and treatment of individuals with a history of mTBI.

Advancement of Technology: NeuroTracker is a state-of-the-art technology which shows promise as a functional biomarker of brain-health, as well as cognitive training tool. NeuroTracker has the ability to serve as an accessible detection method and therapeutic for adults at risk of dementia due to a history of concussion.

Objectives & Experimental Approach: The goal of this research project will be to examine aging older adult males and females with a history of concussion to determine if there are biomarkers that are indicative of cognitive trajectories.

Aim 1 will investigate cognitive-differences in individuals with a history of concussion. The investigators will examine the results of comprehensive neuropsychological and NeuroTracker assessments and task-based neurocognitive performance in older adults (60+ years) with and without histories of concussion.

Aim 2 will identify unique biomarkers from individuals with a history of concussion. The investigators will examine neuroimaging metrics, biomarkers obtained from blood samples, and NeuroTracker performance metrics from older males and females with and without a history of concussion. These results will be compared with those from Aim 1 to help identify positive and negative prognostic predictors for cognitive performance.

Aim 3 will examine how cognitive training with NeuroTracker affects trajectories of aging over time with two longitudinal follow up sessions. Participants will be assigned into a NeuroTracker training, or activities as a normal six-month intervention. The investigators will collect neuropsychological, blood, and neuroimaging biomarkers immediately post-intervention and six-month follow-up time points. Longitudinal follow-up will allow us to examine different trajectories of aging between groups of older adults with and without history of concussion.

Preliminary data: Our preliminary data suggest that adults with and without histories of concussion perform differently on NeuroTracker, and have different neuroimaging signatures. The investigators expect that combining these biomarkers with blood biomarkers will allow for the most comprehensive assessment of brain-health in adults with histories of concussion. NeuroTracker training is an effective cognitive training tool. The investigators expect that 6-months of NeuroTracker intervention will improve brain-health related outcomes in adults aged 60+.

Project Milestones: At the conclusion of year 1 of funding, The investigators expect to have completed participant recruitment and baseline assessments, allowing us to prepare manuscripts based on cross-sectional data from aims 1&2. Year 2 will involve ongoing data analysis with participant follow-ups post-intervention & 6-month follow up, and presentation of initial findings. Year 3 will comprise finishing data collection, presenting longitudinal data and preparing the final manuscript.

Development: Correlations between NeuroTracker baselines and blood biomarker and DTI imaging assessments of brain condition, and correlations between NeuroTracker learning rates with training over time and corresponding improvements in blood biomarker and DTI imaging assessments of brain condition will allow NeuroTracker to market itself as a competitive and accessible health tool.

Deliverables This project is expected to produce definitive correlational data between NeuroTracker, blood-based biomarkers and diffusion tension imaging assessments, establishing combined baselines with unprecedented sensitivity for diagnosing the neurological deficits in aging, caused by a history of concussion. This will establish the relevance of NeuroTracker baselines as a functional biomarker of these long-term effects on brain functioning and brain health, and determine the appropriate assessment protocol for such sensitivity. Additionally, the long-term effects of concussions will be revealed in terms of specific sex and gender differences. Finally, if NeuroTracker is effective at recovering associated neurological deficits, a 6-month bi-weekly training protocol will be validated as a therapeutic intervention, with measures of specifically rejuvenated cognitive functions via standardised neuropsychological assessments. Our team expects to prepare two-academic manuscripts & multiple community presentations (in English and French) to disseminate the results of this study.

Problem Statement and Background Older adults with a history of concussions have a 2x greater risk of developing dementia however it is not clear why some individuals show resilience and are cognitively healthy, while others struggle and show more pronounced cognitive deficits. The sequelae can include physical complaints (e.g. headache, dizziness, nausea, sleep disturbance), cognitive signs (e.g. changes in memory and executive functions), and emotional symptoms (e.g. changes in mood). Although many individuals recover from these symptoms within 10 days, there is now considerable evidence that concussions are a risk factor for the development of neurodegenerative diseases.

Technology Inclusion & Goals NeuroTracker has the potential to serve as a new functional biomarker of brain health and as a cognitive enhancer. It's a task that engages multiple brain networks all at once, demanding the utilization of working memory, complex motion comprehension, and wide-ranging attention management to keep track of numerous objects over time and space. The investigators anticipate that NeuroTracker will synergistically augment the exploratory assessments of long-term concussion effects that rely on blood-based biomarkers and neuroimaging. This unique enhancement could, for the first time, significantly boost the detection sensitivity. Such improvement could reach a level high enough to identify the subtle, yet impactful long-term effects of concussions which may extend into later life. Moreover, this project aims to determine the healing potential of NeuroTracker, specifically as a proactive training tool for cognitive function rehabilitation. This could be pivotal in fostering healthy active aging, allowing individuals to recover and reintegrate cognitive abilities necessary for a vibrant life in their later years.

Research Team: The investigators have assembled a cross-province, diverse multidisciplinary team of experts, allowing us to incorporate state-of-the-art cognitive performance software (i.e. NeuroTracker), neuropsychological assessment, neuroimaging (diffusion tensor imaging; DTI), and blood-based biomarkers, to provide a detailed multimodal framework for assessing the impact of previous concussions. The investigators have also built strong relationships with the Institute for Aging and Life Long Health, as well as the Victoria Brain Injury Society. Our team will have a focus on looking at brain imaging and blood biomarkers, with concurrent neuropsychological and NeuroTracker assessments, and work with graduate and medical school trainees recruited specifically for this project. The identification of biomarkers, including NeuroTracker performance, provides critical insight, as cognitive performance can remain within normal limits when biomarkers of neurodegeneration are present. This is also a critical time-point for interventions aimed at preventing cognitive decline to be instigated. The approaches developed here will be shared within the health care system, both nationally and internationally, given the composition of our team.

Preliminary Data in relation to specific aims: The investigators have recently published several papers that demonstrate our use of neuropsychological assessment and NeuroTracker in elderly and concussed populations; our ability to perform DTI in these populations. Most recently, the investigators have collected preliminary data with 16 participants with a history of concussion and 18 matched controls to examine the extent to which cognitive performance differs between adults with and without a history of concussion. This study examined NeuroTracker performance, as well as cognitive performance using a series of standardized neuropsychological assessments focused on memory, executive functioning, and symptoms of concussion. The results indicated that individuals with remote histories of multiple concussions continue to experience concussion-related symptoms, even years after their injuries (as measured by the Sport Concussion Assessment Tool) and that these individuals had poorer performance across neuropsychological measures of memory and executive functioning. Data from NeuroTracker suggested that individuals with a history of concussion have slower learning curves and worse performance over time than those without.

The investigators have also collected MRI data on older adults with and without a history of concussion, locally at West Coast Medical Imaging (analyses currently in progress), and have completed projects examining diffusion tensor imaging metrics in individuals with dementia compared to healthy controls. Interestingly, another study compared individuals from the Baltimore Longitudinal Study of Aging who reported a concussion an average of 23 years prior, to individuals with no history of concussion, and found that those with prior concussion had microstructural differences in the fornix, anterior corona radiata and superior longitudinal fasciculus using diffusion tensor imaging. They concluded that concussions can produce lasting structural changes in the brain. The proposed study would build on this work by expanding the methods used and investigating longitudinal trajectories.

Methods General Methods and Timelines: A total of 100 aged (60+) adults with a history of concussion and 100 aged adults without a history of concussion will be recruited to the study. Please note that recruitment will be rolling and is anticipated to be complete by year 1.5 of our 3-year timeframe.

The investigators will recruit participants through collaboration with the University of Victoria's Institute on Aging and Lifelong Health, the Victoria Brain Injury Society (VBIS), local media outlets, posters in community spaces, and by word of mouth. A power analysis (GPower Statistical Software) indicates the proposed sample size would be sufficient to determine, at minimum, a moderately weak effect size (f = 0.17). The investigators have chosen to recruit 100 participants per group to account for a maximum of 15% participant attrition over the study period. The sample size is also notably large for a neuroimaging study.

Inclusion criteria will be based on age (60+ years) and history of concussion (with the most recent concussion occurring at least one year prior to the study). Consistent with the literature, the history of concussion will be determined by interviewing participants about their experience with each experience of concussion (e.g. how was the injury sustained (sports injury, vehicle accident, etc.), how long has it been since the injury, did they experience a loss of consciousness during the event, how was their concussion diagnosed, what were their symptoms and when did the symptoms resolve).

The interview will also gather information on age, sex, gender, education, occupation, and medical history (e.g. mood, medications). These variables will be coded and included in analyses, as appropriate. For example, years of education and years since the most recent concussion can be used as covariates. Exclusion criteria include the presence of a diagnosed neurological disorder (e.g. Mild Cognitive Impairment, Alzheimer's disease, Parkinson's disease), history of severe psychiatric disorder (e.g. schizophrenia), or any condition or medication that could affect cognition (e.g. psychotropic, anticholinergic drugs). Exclusion criteria also screen out the presence of any diagnosed visual impairment that could impede NeuroTracker training (i.e. severe colour blindness, monocular vision, blindness), and contraindications for MRI (e.g. metal implants).

Pre-study: A pre-study interview will first determine eligibility for the study, and depending on the preference of the participant, will occur using a either a virtual online meeting platform (Zoom) or as an in-person meeting. If eligible, the research assistant will read the participant consent form with the participant. If the participant provides consent, the research assistant will conduct an intake interview to collect pertinent background information.

Baseline: Participants will complete a comprehensive neuropsychological and NeuroTracker assessment (AIM 1), magnetic resonance imaging (diffusion tensor imaging; DTI) of the brain, and blood collection (AIM 2). Analyses will compare groups with and without a history of concussion as a function of sex and gender.

Intervention: A 6-month intervention will investigate the effects of bi-weekly cognitive training with NeuroTracker, participants with and without histories of concussion will be assigned to either a NeuroTracker intervention or a control (activities as normal) group (balancing for sex/gender).

Follow up: The baseline testing protocol will be repeated for all (200) participants post intervention (Baseline + 6 months) and 6 months (Baseline + one year) follow up. Analyses will examine changes in cognitive scores, blood and neuroimaging biomarkers over time in each group.

Aim 1. Neuropsychological/NeuroTracker methods Aim 1 will investigate differences between older adults with remote histories of concussion and controls using neuropsychological assessment and perceptual-cognitive testing (NeuroTracker). Here the investigators will determine if there are significant differences in cognition (neuropsychological assessment scores) and NeuroTracker assessment scores between individuals with and without prior mTBI. The investigators hypothesize that it will be detected lower cognitive performance in individuals with prior mTBI compared to those without a history of mTBI.

Neuropsychological Assessment Rationale. Neuropsychological assessment is the gold-standard for assessing cognitive performance across domains of function in patients with neurological conditions (including diagnosis of dementia). Many studies use broad screening measures that are less sensitive to the effects of concussion, although it is most common for individuals with mTBI to experience changes in memory, executive function, and mood. For this the investigators will use a more comprehensive approach to neuropsychological assessment with a focus on the following cognitive domains.

NeuroTracker Testing Rationale. NeuroTracker is a perceptual-cognitive task that stimulates multiple brain networks simultaneously, requiring the integration of working memory, complex motion integration, and distributed attention processing to track multiple objects in time and space. Tracking multiple moving objects in three-dimensional space engages many of the same cognitive processes that are affected by concussion, with prior research demonstrating that tests of NeuroTracker may be sensitive to changes after a brain injury has occurred. The investigators have recently shown that NeuroTracker scores can predict cognitive and concussion status in individuals 35 years of age and older, even when the concussion occurred months or years previously. Notably, NeuroTracker training has a robust perceptual component that elicits the integration of several cognitive skills (e.g. processing speed, working memory, visuospatial skills) that 'exercise' the brain more significantly other cognitive tasks (which tend to focus on one cognitive skill, such as memory). As a result, NeuroTracker has significant promise as a functional biomarker for cognitive status in individuals with a history of concussion.

Aim 2. Multimodal biomarker assessment methods Aim 2 will determine if DTI and blood analyses can be used to determine predictive biomarkers for cognitive health in individuals with a history of concussion. These studies will determine if there are significant differences in DTI metrics between individuals with and without prior mTBI. Simultaneously, the investigators will examine if there are significant differences in blood-based biomarkers between individuals with and without prior mTBI, giving us a unique multimodal perspective. The investigators hypothesize that it will be detected specific regions of the brain with decreased white matter integrity (as measured by DTI metrics), increased neuroinflammation, and oxidative stress (as evidenced by blood biomarkers) in individuals with prior mTBI compared to those without a history of mTBI.

Diffusion Tensor Imaging (DTI) Rationale. Magnetic resonance imaging acquisition and post-processing have allowed for diffusion tensor imaging (DTI) based measurements of mean diffusivity and fractional anisotropy, which are indicators of white matter integrity in the brain at a microstructural level. Evidence emerging from DTI research has revealed that individuals with a history of concussion have localized decreases in white matter integrity. For example, a landmark study showed significant changes in DTI metrics in retired NFL players who had sustained multiple concussions compared to matched controls. These individuals also had markedly decreased scores on cognitive measures and higher scores on indices of depression. Other studies replicated these findings in former hockey players who had experienced concussions; they concluded that "advancing age in retired athletes presenting with a history of sports-related concussions is linked to diffuse white matter abnormalities that are consistent with the effects of traumatic axonal injury and exacerbated demyelination." Other studies that have focused on the acute impacts of concussion (before and after hockey season) found significant differences between the sexes, wherein decreased white matter integrity within the superior longitudinal fasciculus, internal capsule, and the corona radiata was found specifically in females and not males. An important next step in this work will be to examine a community-based sample of older female adults with history of concussion (resulting from a mix of etiologies) to determine differences in white matter integrity. It will also be important to link these findings to measures of cognition, emotional well-being (e.g. depression) and other biomarkers, such as blood-based measures. MRI Data collection. Data will be acquired at the West Coast Medical Imaging (WCMI) facility located in Victoria, BC. WCMI has a 3T GE MRI Signa Pioneer Scanner with the ability to collect DTI and high-resolution anatomical data. Structural T1 images will be collected in sagittal orientation with the 3D BRAVO sequence (TR = 8600 ms, TE = 3300 ms, 194 slices, FOV: 256 x 256, voxel size 1 x 1 x 1 mm). T2-weighted fluid-attenuated inversion recovery (FLAIR) images will be obtained for the purpose of WMH volume computation (5.0 mm slice thickness, TE of 90 ms, TR of 945 ms, an inversion time of 2,279 ms, flip angle of 111°, and an in-plane acquisition matrix of 256 x 256). Diffusion tensor imaging data will be collected (axial EPI acquisition with TR = 8000 ms, TE = 101 ms, 52 slices, voxels = 5 x 5 x 2 mm). The scanning protocol will take approximately 30 minutes per participant. The imaging protocol will be followed at baseline and post-intervention & 6-month follow up.

Blood Analysis Rationale. Blood-based protein biomarkers hold particular promise for diagnosing mTBI. Despite evidence that other pathophysiological changes, such as neuroinflammation, oxidative stress, and vascular disruption are prominent, if not universal, features of mTBI neurobiology, virtually no studies have investigated molecules associated with processes outside of neuronal and axonal injury as mTBI biomarkers. One potential biomarker is to assess telomere length. Telomeres are repetitive non-coding DNA sequences located at the end of linear eukaryotic chromosomes, and telomere length is responsive to environmental stressors such as aging (i.e. a marker of cellular senescence), brain injury, and neurodegenerative disease. Blood biomarker quantification: 30mL of whole blood will be collected using standard phlebotomy procedures into BD Vacutainers specific for serum isolation. Dr. Christie has established this procedure at UVic and has appropriate ethical and biosafety certification. Trainee Snowden is a certified phlebotomist with experience in blood draws from elderly participants. Tubes containing blood samples are centrifuged, and the serum is isolated and transferred into .2ml aliquots, flash frozen using liquid nitrogen, and stored at -80°C. Samples are couriered on dry ice to Dr. Shultz's laboratory at Vancouver Island University (Nanaimo) for analysis. Blood protein biomarkers sensitive to pathophysiological processes reflective of neurodegeneration (i.e., p-tau-181), neuroaxonal injury (i.e., NfL, tau, UCHL1), astroglia damage (GFAP), inflammation (e.g., IFNγ, IL-1β, IL-4, IL-5, IL-6, IL-8, IL-10, IL-IL-12p70, IL-17A, IL-18, IL-22, TNFα, C-reactive protein, MMP9), oxidative stress (e.g., 4-HNE, HIF-1), vascular injury (i.e., VEGF, claudin-5, occludin, vWF), and neurotrophic imbalance (i.e., BDNF). Protein biomarkers will be analysed with either the SIMOA HD-X Analyzer or the MesoScale Discovery Quickplex SQ 120. The SIMOA is an advanced digital multiplex ELISA technology platform that offers clinical grade protein biomarker assays. The MesoScale is another sensitive and high-throughput device that allows for testing of more exploratory biomarkers that are not offered on the SIMOA system. By using both devices, the investigators achieve a balance between testing markers ready for clinical use on the SIMOA (i.e., Nf-L, GFAP, UCH-L1, Tau, p-tau-181) and discovering additional markers (e.g., inflammatory cytokines, neurotrophic factors, cerebrovascular injury) with the MesoScale that could be then be developed for clinical application in the case of positive findings. For telomeres, genomic DNA will be extracted from whole-blood and TL will be analyzed with qRT-PCR. At the same time as the blood data collection, a saliva sample will be collected and analyzed to document APOE e status (given that APOE e4 status is a risk factor for Alzheimer's disease and APOE e2 status may be protective).

Aim 3: Intervention with NeuroTracker training Aim 3 of the project is to determine the effectiveness of NeuroTracker for treating cognitive deficits associated with a prior history of concussion.

Intervention Rationale. Dynamic visual attention, or when the brain is called to allocate attention to moving objects, requires perceptual and cognitive skills that are highly called upon in daily life. This type of perceptual-cognitive ability requires higher level processing of complex visual information, reflecting the brain's capacity for integrated functioning. Members of our team have demonstrated that it is possible to train dynamic visual attention in young and older healthy individuals, that the learning trajectory observed during this type of training is highly predictable as well as reproducible, and that gains made during training transfer to athletic performance, to other perceptual skills such as biological motion, and to cognitive function. Moreover, it has also been shown that cerebral resting state changes (captured by qEEG) as a function of training are positively influenced throughout the brain. These changes provide evidence for the power of NeuroTracker to stimulate cerebral plasticity, and suggest that it could facilitate brain reorganization, even years after an injury.

NeuroTracker Intervention Methods. NeuroTracker Core mode will be used to assess the perceptual-cognitive state of each participant. NeuroTracker has a virtual cloud-based platform (NeuroTrackerX), which has been validated for use in research. This online platform allows participants to complete the interventions from home and greatly increases the accessibility of the program. Participants will have two 30-minute training sessions per week over the course of the 6-month intervention. Each session will consist of 3 blocks of 20 trials. For each trial in a block, participants sit upright, approximately 20" away from a standard computer or laptop screen, and wear anaglyph 3D glasses while focusing on the center of a standard 20" computer screen. First, participants are presented with 8 identical yellow balls randomly placed in 3D space on screen.

Second, to identify the necessary targets to be followed, 4 of the balls are briefly highlighted in orange with a white halo. Then, the highlighted balls returned to their original yellow color and begin bouncing within the 3D environment for 8 seconds, after which they are immobilized and the subject is asked to identify the new location of their original target balls. Prior to trial completion, the participant is shown the correct target balls originally highlighted, and the speed of the balls is adjusted in the following trial using a 1-up 1-down staircase procedure. If participants track all 4 balls correctly within a trial, the ensuing trial's ball-bouncing speed is accelerated, and the difficulty continues to increase logarithmically across trials until the participant makes an error, at which point the ball-bouncing speed is reduced in the subsequent trial. This procedure will be done to find the NeuroTracker speed threshold criterion at which the participant could correctly identify all of the targets 50% of the time, i.e. the point at which their performance neither improved, nor deteriorated. The mean speed threshold across all 3 testing blocks, is calculated automatically by the NeuroTracker Core program, will be used as a measure of performance, wherein higher NeuroTracker scores indicate higher perceptual-cognitive abilities.

Post-intervention and 6-Month Follow up. Following the NeuroTracker intervention and at 6-month follow up, data collection will include neuroimaging, blood collection, neuropsychological assessment and a single NeuroTracker session, using the methods described under Aim 1.

Project Management Plan: The research team acknowledges the scope of this project, and has developed a preliminary project management plan to ensure the feasibility of the project. In the budget, the investigators have accounted for two full-time research coordinators (one at UdeM, one at UVic) to facilitate this project. In addition, he investigators will have two full time graduate students, one full-time research assistant and three honours students directly working on this project. The team will meet virtually once per month to provide updates and build plans.

ELIGIBILITY:
Inclusion Criteria:

* It will be based on age (60+ years) and history of concussion (with the most recent concussion occurring at least one year prior to the study). Consistent with the literature, the history of concussion will be determined by interviewing participants about their experience with each experience of concussion (e.g. how was the injury sustained (sports injury, vehicle accident, etc.), how long has it been since the injury, did they experience a loss of consciousness during the event, how was their concussion diagnosed, what were their symptoms and when did the symptoms resolve).

The interview will also gather information on age, sex, gender, education, occupation, and medical history (e.g. mood, medications). These variables will be coded and included in analyses, as appropriate. For example, years of education and years since the most recent concussion can be used as covariates.

Exclusion Criteria:

* Include the presence of a diagnosed neurological disorder (e.g. Mild Cognitive Impairment, Alzheimer's disease, Parkinson's disease), history of severe psychiatric disorder (e.g. schizophrenia), or any condition or medication that could affect cognition (e.g. psychotropic, anticholinergic drugs). Exclusion criteria also screen out the presence of any diagnosed visual impairment that could impede NeuroTracker training (i.e. severe colour blindness, monocular vision, blindness), and contraindications for MRI (e.g. metal implants).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological cognitive assessments | By the end of the second year.
  Changes from Baseline, follow-up 1 (3 months), and follow-up 2 (6 months) on: 1) the Verbal Fluency Score (number of words, standardized Z-score) as assessed by the Verbal Fluency Test (FAS & Animals).
Neuropsychological cognitive assessments | By the end of the second year.
  Changes from Baseline, follow-up 1 (3 months), and follow-up 2 (6 months) on: 2) The Verbal Learning and Memory Score (the number of words recalled, standardized Z-score) as assessed by the California Verbal Learning Test - Second Edition (CVLT-II), with the alternate version used for follow-ups.
Neuropsychological cognitive assessments | By the end of the second year.
  Changes from Baseline, follow-up 1 (3 months), and follow-up 2 (6 months) on:
  3) The Processing Speed Score (number of correct responses, standardized Z-score) as assessed by the Symbol Digit Modalities Test.
Neuropsychological cognitive assessments | By the end of the second year.
  Changes from Baseline, follow-up 1 (3 months), and follow-up 2 (6 months) on: 4) The Working Memory Score (total correct sequences, standardized Z score), as assessed by the Digit Span (forward, backward, sequencing).
Neuropsychological cognitive assessments | By the end of the second year.
  Changes from Baseline, follow-up 1 (3 months), and follow-up 2 (6 months) on: 5) The Executive Function Score (Time in seconds, Number of errors, Standardized Z scores) as assessed by the Trail Making Test A & B.
Neuropsychological cognitive assessments | By the end of the second year.
  Changes from Baseline, follow-up 1 (3 months), and follow-up 2 (6 months) on: 6) The Global Cognitive Function Score (Total score, 0-30) as evaluated by the Mini-Mental State Exam (MMSE).
Multimodal biomarker assessment | By the end of the second year
  Changes from Baseline, follow-up 1 (3 months), and follow-up 2 (6 months) on: 1) the Fractional Anisotropy (FA) in A Priori ROIs (Unitless) as evaluated by Diffusion Tensor Imaging (DTI).
Multimodal biomarker assessment | By the end of the second year
  Changes from Baseline, follow-up 1 (3 months), and follow-up 2 (6 months) on: 2) The Mean Diffusivity in A Priori ROIs (mm2/s) as evaluated by Diffusion Tensor Imaging (DTI).
Multimodal biomarker assessment | By the end of the second year
  Changes from Baseline, follow-up 1 (3 months), and follow-up 2 (6 months) on: 3) The Number of Clusters With Group Differences in FA (number of clusters) as evaluated by Diffusion Tensor Imaging (DTI).
Multimodal biomarker assessment | By the end of the second year
  Changes from Baseline, follow-up 1 (3 months), and follow-up 2 (6 months) on: 4) The Number of Clusters With Group Differences in MD (number of clusters) as evaluated by Diffusion Tensor Imaging (DTI).
NeutroTracker assessement | By the end of the second year
  Changes from Baseline, follow-up 1 (3 months), and follow-up 2 (6 months) on the Perceptual-Cognitive Tracking Score (Speed threshold, arbitrary units) as evaluated by NeuroTracker.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Faubert Principal Investigator, PhD, Principal Investigator — Université de Montréal
Locations (3):
- Canada (3):
  - Christie Lab, Victoria, British Columbia
  - Jodie Gawryluk, Victoria, British Columbia
  - Faubert Lab, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Use of the wii balance board to assess changes in postural balance across athletic season HM Cullen, Y Sun, BR Christie, EP Zehr British Journal of Sports Medicine 51 (11), A1-A1
- [Background] Relationship between king devick TEST, SCAR3 and 3D mot in cognitive assessment KR Oslund, HM Cullen, K Kowalski, B Christie British Journal of Sports Medicine 51 (11), A9-A10
- [Background] Three-Dimensional Multiple Object Tracking as A Marker of Normal Cerebral Functioning after Paediatric Mild Traumatic Brain Injury: A Pilot Study LA Corbin-Berrigan, K Kowalski, J Faubert, B Christie, I Gagnon BRAIN INJURY 33, 137-138
- [Background] 3-Dimensional Multiple Object Tracking Training Can Enhance Selective Attention, Psychomotor Speed, and Cognitive Flexibility in Healthy Older Adults CR Spaner, S Musteata, RA Kenny, JR Gawryluk, S Hofer, BR Christie Ageing Science and Mental Health Studies 3 (4), 1-12
- [Background] A pilot study of diffusion tensor imaging metrics and cognitive performance pre and post repetitive, intentional sub-concussive heading in soccer practice RA Kenny, CD Mayo, S Kennedy, AA Varga, L Stuart-Hill, ...Journal of Concussion 3, 2059700219885503
- [Background] Perceptual-Cognitive Training Can Improve Cognition in Older Adults with Subjective Cognitive Decline CBR Musteata Stella, Yoshida Kaya, Baranzini Daniele, Spaner Caroline ... Ageing Science and Mental Health Studies 3 (6), 1-15
- [Background] Effects of 3D-Multiple Object Tracking on Reaction Time Performance in High-Performance Varsity Swimmers TM Snowden, KC Hogan, TJ Sparks, RG Stein, LM Melanie R, BR Christie Journal of Athletic Enhancement 9 (1), 1-12
- [Background] Corbin-Berrigan LA, Kowalski K, Faubert J, Christie B, Gagnon I. Could Neurotracker be used as a clinical marker of recovery following pediatric mild traumatic brain injury? An exploratory study. Brain Inj. 2020 Feb 23;34(3):385-389. doi: 10.1080/02699052.2020.1723699. Epub 2020 Feb 4. PMID 32013583
- [Background] Lysenko-Martin MR, Hutton CP, Sparks T, Snowden T, Christie BR. Multiple Object Tracking Scores Predict Post-Concussion Status Years after Mild Traumatic Brain Injury. J Neurotrauma. 2020 Aug 15;37(16):1777-1787. doi: 10.1089/neu.2019.6842. Epub 2020 Apr 17. PMID 31950862
- [Background] Cavanagh P, Alvarez GA. Tracking multiple targets with multifocal attention. Trends Cogn Sci. 2005 Jul;9(7):349-54. doi: 10.1016/j.tics.2005.05.009. PMID 15953754
- [Background] Manley G, Gardner AJ, Schneider KJ, Guskiewicz KM, Bailes J, Cantu RC, Castellani RJ, Turner M, Jordan BD, Randolph C, Dvorak J, Hayden KA, Tator CH, McCrory P, Iverson GL. A systematic review of potential long-term effects of sport-related concussion. Br J Sports Med. 2017 Jun;51(12):969-977. doi: 10.1136/bjsports-2017-097791. Epub 2017 Apr 28. PMID 28455362
- [Background] Do sub-concussive impacts from soccer heading in practice cause changes in brain structure and function? (2018-09-11) Kenny, Rebecca; Christie, Brian R.; Gawryluk, Jodie R. Thesis. University of Victoria.
- [Background] Snowden T, Ohlhauser L, Morrison J, Faubert J, Gawryluk J, Christie BR. A Protocol for Remote Cognitive Training Developed for Use in Clinical Populations During the COVID-19 Pandemic. Neurotrauma Rep. 2023 Aug 14;4(1):522-532. doi: 10.1089/neur.2023.0009. eCollection 2023. PMID 37645472
- See also: Principal Investigator website — http://faubertlab.com/